CLINICAL TRIAL: NCT00579735
Title: Histologic Diagnoses of Incidentally Detected Lesions on MRI
Status: Withdrawn | Type: Observational
Why Stopped: No subjects were ever enrolled. This study was closed at the IRB.
Sponsor: University of Arkansas (Other)
Responsible Party: Steven E. Harms, MD, UAMS
Other Study IDs: 37640
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients who received breast MRI will be evaluated for a variety of indications including : # each indication : 1) known cancer staging for local exent, 2)high risk, 3)high suspicion clinical finding, 4)questionable mammo finding, 5)silicone leak The number of incidental lesions not detected by any other method that were subsequently subjected to biopsy with the following BIRADS categories 3-# reasons for bx 4-# 5-# Of the lesions detected % of each BIRADS category were postive histologies-ductal, lobular, DCIS, etc. and negative (fibrosis, hyperplasia, etc.) Criteria for classification: morphology, dynamics, clinical significance will be evaluated and a predictive value established.

DETAILED DESCRIPTION:
Patients who received breast MRI will be evaluated for a variety of indications including ? # each indication : 1) known cancer staging for local exent, 2)high risk, 3)high suspicion clinical finding, 4)questionable mammo finding, 5)silicone leak The number of incidental lesions not detected by any other method that were subsequently subjected to biopsy with the following BIRADS categories 3-# reasons for bx 4-# 5-# Of the lesions detected % of each BIRADS category were postive histologies-ductal, lobular, DCIS, etc. and negative (fibrosis, hyperplasia, etc.) Criteria for classification: morphology, dynamics, clinical significance will be evaluated and a predictive value established. This study is limited to retrospective chart review with the only foreseeable risk being that of disclosure of PHI. To minimize this risk, data collection forms will be identified by subject ID number. A master list of these ID numbers linked to subject medical record number will be maintained in the investigator's file and kept in a secure location accessible only to the study team for purposes of verification of data and validation of results. The medical record number will not be recorded on any other form containing subject PHI. The only foreseeable breach of confidentiality would be for the security of the investigator's files to be compromised

ELIGIBILITY:
Inclusion Criteria:

* All patients subjected to biopsy as a result of findings seen only on MRI

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mammography clinic in Northwest Arkansas
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Harms, MD, Principal Investigator — University of Arkansas